CLINICAL TRIAL: NCT05891041
Title: First Study: InterPoc's Safety and Tolerability in Adults With Second Study: Safety and Functionality of InterPoc
Brief Title: New Method for the Collection of the Output From the Ileostoma Using a Intestinal Tampon
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Patrick Achiam, DMSCI, associate professor, Rigshospitalet, Denmark
Other Study IDs: H-23000001
Record Dates: First submitted 2023-05-01; First posted 2023-06-06 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1 study: A pilot study of 8 adults with ileostomy was included in this trial of "first in human" with InterPoc™, an absorbent intestinal tampon safety and feasibility in humans with ileostomies.

Study 2: A study in total with 24 participants, evaluating both the safety but also the functionality of InterPoc in humans with ileostomies.

DETAILED DESCRIPTION:
Approximately 1 million individuals with ileostomies face limitations in design and complications with traditional stoma bags dating back to the 1950s. Colostomy care alternatives are unavailable for ileostomy patients, prompting the development of InterPoc™, an absorbent intestinal tampon.

The first study aims to assess its safety and feasibility in humans, while the second study focuses of the overall safety and functionality of the tampon in all 24 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 Ileostoma at least created 6 months prior Ileostoma opening of at least 15 mm

Exclusion Criteria:

Inflamatory condition in the stoma or other intestine diagnosed within 2 months of the study Parastomal hernia daily output above 2 litters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients with an ileostoma
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of patients requiring pharmacological or surgical intervention due to the use of InterPOC for 6 hours | 6 hours
  Safety of Interpoc during use

SECONDARY OUTCOMES:
Pain during interpoc use | 6 hours
  Using the NRS from 0-10
Early warning score during interpoc use (vital signs Pulse, blood pressure, oxygen saturation, respiratory rate, temperature), | 6 hours
  A low score is better than a high score
Scale (0-10) score of Discomfort, acid reflux, nausea | 6 hours
  A low score is better than a high score
InterPoc™ weight before and after insertion | 6 hours
  For comparable
Leakage around the stoma pouch | 6 hours
  Scale: 1-3)
Fecal output in stoma bag (ml) before and after the trail | 6 hours
  scale 1-3
InterPoc™ Skin Irritation | 6 hour
  (Scale: 1-3)
Insertion and removal resistance | 6 hour
  scale 1-3)
Food consumption | 6 hour
  descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, København Ø, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No